CLINICAL TRIAL: NCT05284474
Title: Management of Early-onset Fetal Growth Restriction: Angiogenic Factors Versus Feto-placental Doppler (Early GRAFD)
Brief Title: Management of Early-onset Fetal Growth Restriction: Angiogenic Factors Versus Feto-placental Doppler
Acronym: earlyGRAFD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PR(AMI)113/2022
Record Dates: First submitted 2022-02-13; First posted 2022-03-17 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Fetal Growth Retardation; Preeclampsia; Placenta Diseases
Keywords: fetal growth restriction; small for gestational age; PlGF; sFlt-1; Doppler
MeSH Terms: conditions — Fetal Growth Retardation; Pre-Eclampsia; Placenta Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Small fetuses will be classified into 5 severity stages and managed as follows:
  * SGA: Estimated fetal weight (EFW) between p3 and p10 with normal Dopplers. Ultrasound/2 weeks, elective vaginal delivery at ≥39-40 weeks.
  * Stage I: EFW ≤p3 p or EFW p3-10 + UA PI >p95 and/or UtA PI >p95, and, at ≥32 weeks, CPR and/or MCA PI <p5, in 2 occasions >12 hours apart. Ultrasound weekly, elective vaginal delivery at ≥37 weeks.
  * Stage II: AEDF UA in 2 occasions >12 hours apart. Ultrasound every 48-72h, elective Cesarean delivery at ≥34 weeks.
  * Stage III: DV PI > p95 (or absent DV "a" wave) or reversed end-diastolic UA >50% of cycles, in both cases in two occasions > 6 hours apart. Ultrasound every 24-48h, elective Cesarean delivery at ≥30 weeks.
  * Stage IV: reversed DV "a" wave in two occasions > 6 hours apart. Elective Cesarean delivery at ≥26 weeks.
- Study (Experimental): Doppler protocol (as in controls) + sFlt-1/PlGF ratio cutoffs will be incorporated as follows:
  * <38: Ultrasound biweekly in stage I FGR and every four weeks in SGA. In both cases delivery at ≥39-40 weeks.
  * 38-110: In stage I FGR and SGA ultrasound weekly. Delivery at ≥37 weeks.
  * >110: In stage I FGR and SGA ultrasound weekly. Delivery at ≥36 weeks.
  * >110 and concurrent preeclampsia: In stage I FGR and SGA ultrasound every 48h-72h. Delivery at ≥34 weeks.
  * >201: Ultrasound every 48-72h, delivery at ≥34+0 weeks. If concurrent preeclampsia, delivery at ≥32+0 weeks.
  * >655: Ultrasound every 48-72h, delivery at ≥32+0 weeks. If concurrent preeclampsia, delivery at ≥30+0 weeks.
  * >1000: In cases with concurrent PE, delivery at ≥29+0 weeks.
  Interventions: Diagnostic Test: soluble fms-like tyrosine kinase to placental growth factor ratio (sFlt-1/PlGF)

INTERVENTIONS:
Diagnostic Test: soluble fms-like tyrosine kinase to placental growth factor ratio (sFlt-1/PlGF) — soluble fms-like tyrosine kinase to placental growth factor ratio (sFlt-1/PlGF) will be incorporated to the management of early-onset small fetuses (estimated fetal weight ≤10th percentile)
  Arms: Study

SUMMARY:
This is a multicentre, open-label, randomized controlled trial. A total of 340 singleton pregnancies with an EFW ≤10th percentile between 26+0 and 31+6 weeks will be recruited and randomly allocated to either the control or the intervention group. In the control group, standard Doppler-based management will be used. In the intervention group, different soluble fms-like tyrosine kinase to placental growth factor ratio (sFlt-1/PlGF) cutoffs will be incorporated to the current protocol to adjust the frequency of ultrasounds and to plan elective delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of at least 18 years old
* Singleton pregnancy
* Ultrasonographic EFW ≤10th percentile between 26+0 and 31+6 weeks of gestation
* Gestational age confirmed by fetal crown-rump length measurement during the first trimester scan (from 11+0 to 13+6 weeks of gestation) or by in vitro fertilization dates.

Exclusion Criteria:

* Major fetal malformations or genetic disorders
* Fetal death
* Refusal to give informed consent
* Stage IV FGR

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 340 (Estimated)
Dates: Start 2024-06-03 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Fetal and Neonatal complications | During pregnancy and up to 28 days after delivery
  stillbirth, neonatal death, artery cord pH ≤7.0, respiratory distress syndrome, required invasive ventilatory support, grade III or IV intraventricular hemorrhage, neonatal sepsis, necrotizing enterocolitis, neonatal seizures, pneumonia, meningitis, broncopulmonary dysplasia, hypoxic ischemic encephalopathy, Apgar score <7 at 5 minutes, or elective delivery at <28 weeks of gestation.
Composite adverse maternal outcome | During pregnancy and up to 28 days after delivery
  Progression to PE with severity features; progression to hemolysis, elevated liver enzymes, and low platelet count (HELLP) syndrome (LDH >600 IU/L, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) elevated more than twice the upper limit of normal, and the platelet count less than 100 X 109/L); eclampsia, stroke, hepatic hematoma or rupture; oliguria (urine output of <400 mL during 24 hours, or need for treatment with furosemide to maintain urine output at >400 mL for 24 hours); cardiovascular dysfunction (need for inotropic support, left ventricle failure, or myocardial infarction); placental abruption; maternal death; maternal admission to intensive care unit >48 hours, and/or requirement for blood transfusion.

SECONDARY OUTCOMES:
Maternal perceived stress | At inclusion and 4 weeks later
  Mean and sd or median and IQR of the score obtained in the perceived stress scale in each group
Other perinatal outcomes | During pregnancy and up to 28 days after delivery
  transient tachypnea, non-invasive ventilatory support, hypoglycemia, neonatal jaundice (treated with phototherapy), rate of elective deliveries < 30 weeks, <34 weeks and < 37 weeks for FGR and/or PE, birthweight <3 rd and <10th percentiles, mode of delivery (vaginal, instrumental vaginal delivery and Cesarean), rate of Cesarean delivery for abnormal CTG, median maternal stay in ICU, median neonatal stay in N-ICU, maternal corticosteroids (single dose, complete course), prenatal magnesium sulfate (at least 4h) for preterm delivery.
Number of ultrasounds per participant | During pregnancy (before and after 37 weeks)
  Mean and sd or median and IQR in each group

CONTACTS AND LOCATIONS:
Overall Officials: Manel Mendoza, MD, PhD, Principal Investigator — Vall d'Hebron Institut de Recerca (VHIR)
Locations (27):
- Spain (27):
  - Complejo Hospitalario Universitario de A Coruña, A Coruña
  - Hospital Universitario General de Alicante, Alicante
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Vall d'hebron Barcelona Hospital Campus, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario de Getafe, Getafe
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario San Cecilio, Granada
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Materno Infantil de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitari Son Llàtzer, Palma de Mallorca
  - Corporació Sanitària Parc Taulí, Sabadell
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Virgen de Valme, Seville
  - Virgen Macarena, Seville
  - Hospital Universitario Joan XXIII de Tarragona, Tarragona
  - Consorci Sanitari de Terrassa, Terrassa
  - Hospital Universitari Mútua Terrassa, Terrassa
  - Hospital Universitario de Torrejón, Torrejón de Ardoz
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided